CLINICAL TRIAL: NCT02392000
Title: Mobile Sleep and Pain Intervention for OEF, OIF and OND Veterans
Brief Title: Mobile Sleep Intervention for OEF, OIF and OND Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Rochester (Other); Northeastern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPO 14-144
Record Dates: First submitted 2015-02-12; First posted 2015-03-18 (Estimated); Results first posted 2018-03-09 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-03

CONDITIONS: Chronic Insomnia
Keywords: chronic insomnia; Veterans Health
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- WatchPAT and CBT-i Coach mobile app (Experimental): Individuals use the WatchPAT sleep monitor and the CBT-i Coach app to self-manage insomnia
  Interventions: Device: WatchPAT sleep monitor; Behavioral: CBT-i Coach mobile app

INTERVENTIONS:
Device: WatchPAT sleep monitor — Self-management of insomnia using a mobile sleep device
Behavioral: CBT-i Coach mobile app — Self-management of insomnia using a mobile app based on Cognitive Behavioral Therapy for Insomnia

SUMMARY:
Many Veterans of the recent wars in Iraq and Afghanistan struggle with chronic insomnia (trouble falling or staying asleep). Most current interventions for insomnia are time-consuming, making it difficult for this younger, working group of Veterans to use and benefit from these interventions. The investigators will assess whether Veterans find it helpful to use two health information technology tools, one for measuring participant sleep (the WatchPAT) and one for managing participant sleep (the CBTI Coach). The WatchPAT will measure physiological sleep in the Veteran participant's home. The CBTI Coach is a mobile health application used on the Veteran's mobile phone or tablet to teach skills that can reduce insomnia. The investigators will combine use of the WatchPAT with the CBTI Coach so Veterans can self-manage insomnia at home. Participants will record their physiological sleep and self-report on their sleep at home during a 6 week self-management program. The investigators will measure if Veterans find the tools helpful and easy to use, and which Veterans find the tools most helpful.

DETAILED DESCRIPTION:
Sleep disturbance in the form of chronic insomnia (difficulty in falling or staying asleep) is a major health care problem for Operation Enduring Freedom (OEF), Operation Iraqi Freedom (OIF), and Operation New Dawn (OND) Veterans. Chronic insomnia is often co-morbid with mental and behavioral health issues such as posttraumatic stress disorder (PTSD) and mild traumatic brain injury (mTBI), which are common in these Veterans. Current behavioral interventions like cognitive behavioral therapy for insomnia (CBTI) that are used to treat chronic insomnia are effective, but time-consuming. As a result, this largely younger, working cohort of Veterans does not use and benefit from these interventions as much as they could. The investigators will assess the usability and feasibility of two health information technology (HIT) tools for measuring objective and subjective sleep, and for self-managing chronic insomnia. An existing mobile sleep monitoring device used by some VA sleep clinics, the WatchPAT, will be used to measure objective sleep parameters in the Veteran's home. A benefit of this tool is that it can detect probable sleep apnea, which will permit referral of these Veterans for sleep apnea treatment instead of insomnia self-management. An existing VA mobile health application (or app), the CBTI Coach, can be used on a mobile device to teach skills to reduce insomnia based on the elements of manualized CBTI. The goal is to combine the WatchPAT and the CBTI Coach along with self-management guidance to help Veterans with chronic insomnia learn how to improve their sleep. As part of a 6-week pre-post intervention pilot usability and feasibility trial, patients will record their objective and subjective sleep at home at the beginning of the 6-week self-management trial and again at the end. Subjective sleep reports in the form of sleep diaries will be measured throughout the program as part of using the CBTI Coach app. The objective and subjective sleep reports will be combined and accessible from the mobile device and can be used to help guide sleep self-management by the participant. Self-management will be aided by self-management worksheets and features of the CBTI Coach App. Usability of the two HIT tools will be assessed within the conceptual framework of an Integrated Technology Acceptance Model via survey items about each of the HIT tools. Feasibility will be assessed using measures of the number of times that elements of the CBTI Coach were accessed during the 6-week program, and from a semi-structured qualitative interview conducted at the end of the program. In the interview, the investigators will obtain information about the barriers to and facilitators of use of the WatchPAT and CBTI Coach. If there is high use of these tools for insomnia self-management, then the pilot study will have provided important incremental value to the new VA CBTI Coach app. The investigators also will collect data about the user factors that impact use of the tools (e.g., depression, mild traumatic brain injury, age), and thereby either be able to target the tools toward those most likely to use them, or suggest further developments to increase use by potential users. The pilot sample will provide preliminary data on sleep outcomes. The proposed work is responsive to multiple priority areas for HSR&D including Healthcare Informatics, Healthcare Access, Mental and Behavioral Health, and Post-deployment Health. By partnering with the VA Office of Connected Health (Web and Mobile Solutions), the VA's eHealth QUERI, and the developers of the VA CBTI Coach App, the investigators will ensure that these findings are maximally useful for future versions of the CBTI Coach app. The investigators also will be able to determine the usefulness of an integrated mobile sleep assessment and self-management program that can be used by Veterans anywhere.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have served in the most recent wars in Iraq or Afghanistan (OIF, OEF or OND),
* be age 21-65,
* report current insomnia as defined by an Insomnia Index Severity 40 score > 10 5,79,
* and report insomnia duration of at least 1 month and impaired daytime functioning (as measured by endorsing Much or Very Much on ISI Item 7 about how much sleep problems interfere with daily functioning).
* In addition, eligible individuals must be willing to use a device provided by the study team (an iPod touch).

Exclusion Criteria:

* Exclusions will include self-reported (or in-study determined) sleep apnea that is more than mild,
* periodic leg movements,
* or circadian rhythm disorder (delayed or advanced sleep phase).
* Exclusions for WatchPAT use include use of alpha blockers or short-acting nitrates,
* permanent pacemaker, or
* sustained non-sinus cardiac arrhythmias. Sleep apnea will be assessed from the WatchPAT on the first night of objective sleep testing and participants excluded from further participation if apnea is documented.
* Other exclusions include moderate to severe cognitive impairment defined by scores on the Telephone Mini Mental State Exam,
* inability to speak and read English,
* or malformation of the fingers that would preclude use of the WatchPAT device.
* In addition, individuals meeting criteria for current active psychosis, mania, suicidal ideation with plan and intent, or excessive alcohol use as determined using the AUDIT-C will be excluded from participation.
* Those with greater than mild sleep apnea as determined based on a WatchPAT-based Apnea-Hypopnea Index [AHI] > 15/hour of sleep, will be withdrawn from the study and referred for sleep apnea treatment.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2016-11-16 (Actual); Study Completion 2016-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen S. Quigley, PhD, Principal Investigator — Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA
Locations (1):
- Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA, Bedford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaitz J, Robinson SA, Petrakis BA, Reilly ED, Chamberlin ES, Wiener RS, Quigley KS. Veteran Acceptance of Sleep Health Information Technology: a Mixed-Method Study. J Technol Behav Sci. 2023;8(1):57-68. doi: 10.1007/s41347-022-00287-x. Epub 2022 Dec 13. PMID 36530383
- [Derived] Reilly ED, Robinson SA, Petrakis BA, Kuhn E, Pigeon WR, Wiener RS, McInnes DK, Quigley KS. Mobile App Use for Insomnia Self-Management: Pilot Findings on Sleep Outcomes in Veterans. Interact J Med Res. 2019 Jul 24;8(3):e12408. doi: 10.2196/12408. PMID 31342904

RESULTS

PARTICIPANT FLOW:
Groups:
- WatchPAT and CBT-i Coach App: Individuals use the WatchPAT sleep monitor and the CBT-i Coach app to self-manage insomnia
  WatchPAT sleep monitor: Self-management of insomnia using a mobile sleep device
  CBT-i Coach mobile app: Self-management of insomnia using a mobile app based on Cognitive Behavioral Therapy for Insomnia
Period: Overall Study
Arm/Group | WatchPAT and CBT-i Coach App
Started | 38
Completed | 11
Not Completed | 27
Not completed — Greater than mild sleep apnea exclusion | 18
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 8

BASELINE CHARACTERISTICS:
Arm/Group | WatchPAT and CBT-i Coach App
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 31
  More than one race | 3
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38
Height [Mean (Standard Deviation); unit: inches] | 68.6 (3.8)
Weight [Mean (Standard Deviation); unit: pounds] | 195.9 (40.5)
Usability Satisfaction with Care [Mean (Standard Deviation); unit: units on a scale] — The minimum for this subscale score is 3. The maximum for this subscale score is 21. Higher scores indicate greater satisfaction with their medical care. These scores are from the Usability Survey which is given only at the baseline and used to predict later tech use. Also, because this predictor is measured at baseline to predict initiation of tech use, we can use the complete, enrolled sample of 38, even if individuals are withdrawn later for apnea.
  units on a scale | 14.6 (3.1)
Usability Health Knowledge [Mean (Standard Deviation); unit: units on a scale] — The minimum for this subscale score is 2. The maximum for this subscale score is 14. Higher scores indicate greater health knowledge. These scores are from the Usability Survey which is given only at the baseline and used to predict later tech use. Also, because this predictor is measured at baseline to predict initiation of tech use, we can use the complete, enrolled sample of 38, even if individuals are withdrawn later for apnea.
  units on a scale | 8.0 (2.4)
Usability Internet Dependence [Mean (Standard Deviation); unit: units on a scale] — The minimum for this subscale score is 4. The maximum for this subscale score is 28. Higher scores indicate greater internet dependence. These scores are from the Usability Survey which is given only at the baseline and used to predict later tech use. Also, because this predictor is measured at baseline to predict initiation of tech use, we can use the complete, enrolled sample of 38, even if individuals are withdrawn later for apnea.
  units on a scale | 19.5 (5.6)
Usability Information Seeking Preferences [Mean (Standard Deviation); unit: units on a scale] — The minimum for this subscale score is 4. The maximum for this subscale score is 28. Higher scores indicate greater preference for seeking information. These scores are from the Usability Survey which is given only at the baseline and used to predict later tech use. Also, because this predictor is measured at baseline to predict initiation of tech use, we can use the complete, enrolled sample of 38, even if individuals are withdrawn later for apnea.
  units on a scale | 21.8 (4.4)
Usability Healthcare Need [Mean (Standard Deviation); unit: units on a scale] — The minimum for this subscale score is 0. The maximum for this subscale score is 4. Higher scores indicate greater health care need. These scores are from the Usability Survey which is given only at the baseline and used to predict later tech use. Also, because this predictor is measured at baseline to predict initiation of tech use, we can use the complete, enrolled sample of 38, even if individuals are withdrawn later for apnea.
  units on a scale | 1.3 (1.0)
CBT-i Coach App Intrinsic Motivation [Mean (Standard Deviation); unit: units on a scale] — The minimum for this subscale score is 3. The maximum for this subscale score is 21. Higher scores indicate greater intrinsic motivation to use the CBT-i Coach app. These scores are from the Usability Survey which is given only at the baseline and used to predict later tech use. Also, because this predictor is measured at baseline to predict initiation of tech use, we can use the complete, enrolled sample of 38, even if individuals are withdrawn later for apnea.
  units on a scale | 14.7 (3.2)
CBT-i Coach Perceived Ease of Use [Mean (Standard Deviation); unit: units on a scale] — The minimum for this subscale score is 3. The maximum for this subscale score is 21. Higher scores indicate greater perceived ease of use of the CBT-i Coach app. These scores are from the Usability Survey which is given only at the baseline and used to predict later tech use. Also, because this predictor is measured at baseline to predict initiation of tech use, we can use the complete, enrolled sample of 38, even if individuals are withdrawn later for apnea.
  units on a scale | 16.1 (2.9)
CBT-i Coach Perceived Usefulness [Mean (Standard Deviation); unit: units on a scale] — The minimum for this subscale score is 3. The maximum for this subscale score is 21. Higher scores indicate greater perceived usefulness of the CBT-i Coach app. These scores are from the Usability Survey which is given only at the baseline and used to predict later tech use. Also, because this predictor is measured at baseline to predict initiation of tech use, we can use the complete, enrolled sample of 38, even if individuals are withdrawn later for apnea.
  units on a scale | 15.9 (3.0)
CBT-i Coach Behavioral Intention [Mean (Standard Deviation); unit: units on a scale] — The minimum for this subscale score is 2. The maximum for this subscale score is 14. Higher scores indicate greater behavioral intention to use the CBT-i Coach app. These scores are from the Usability Survey which is given only at the baseline and used to predict later tech use. Also, because this predictor is measured at baseline to predict initiation of tech use, we can use the complete, enrolled sample of 38, even if individuals are withdrawn later for apnea.
  units on a scale | 12.5 (2.1)
WatchPAT Intrinsic Motivation [Mean (Standard Deviation); unit: units on a scale] — The minimum for this subscale score is 3. The maximum for this subscale score is 21. Higher scores indicate greater intrinsic motivation to use the WatchPAT. These scores are from the Usability Survey which is given only at the baseline and used to predict later tech use. Also, because this predictor is measured at baseline to predict initiation of tech use, we can use the complete, enrolled sample of 38, even if individuals are withdrawn later for apnea.
  units on a scale | 13.9 (3.8)
WatchPAT Perceived Ease of Use [Mean (Standard Deviation); unit: units on a scale] — The minimum for this subscale score is 3. The maximum for this subscale score is 21. Higher scores indicate greater perceived ease of use of the WatchPAT. These scores are from the Usability Survey which is given only at the baseline and used to predict later tech use. Also, because this predictor is measured at baseline to predict initiation of tech use, we can use the complete, enrolled sample of 38, even if individuals are withdrawn later for apnea.
  units on a scale | 16.7 (3.4)
WatchPAT Perceived Usefulness [Mean (Standard Deviation); unit: units on a scale] — The minimum for this subscale score is 3. The maximum for this subscale score is 21. Higher scores indicate greater perceived usefulness of the WatchPAT. These scores are from the Usability Survey which is given only at the baseline and used to predict later tech use. Also, because this predictor is measured at baseline to predict initiation of tech use, we can use the complete, enrolled sample of 38, even if individuals are withdrawn later for apnea.
  units on a scale | 16.3 (3.3)
WatchPAT Behavioral Intention [Mean (Standard Deviation); unit: units on a scale] — The minimum for this subscale score is 2. The maximum for this subscale score is 14. Higher scores indicate greater behavioral intention to use the WatchPAT. These scores are from the Usability Survey which is given only at the baseline and used to predict later tech use. Also, because this predictor is measured at baseline to predict initiation of tech use, we can use the complete, enrolled sample of 38, even if individuals are withdrawn later for apnea.
  units on a scale | 12.6 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Using WatchPAT
Description: Use of WatchPAT on 3 nights. In Week 0 it is the number of participants who used the WatchPAT that Week (and participants had two possible nights during that week that they could use the WatchPAT). In Week 6 it is the number of participants who used the WatchPAT that Week (and participants had one night that they could use the WatchPAT). We measured participant adherence using a count of the number of participants who used the WatchPAT at Week 0, and the number of participants using the WatchPAT at Week 6.
Time Frame: Week 0 (Pre-Intervention) and Week 6 (Post-Intervention)
Population: Those who completed enrollment and were not withdrawn by study personnel for insomnia are those whose data are used for Week 0.
Measure: Count of Participants; unit: Participants
Arm/Group | WatchPAT and CBT-i Coach Mobile App
Number analyzed (Participants) | 11
Participants
  Number of Participants using WatchPAT at Baseline | 11
  Number of Participants using WatchPAT at Week 6 | 11

2. Primary Outcome: Number of Participants Using CBT-I Coach
Description: CBT = Cognitive Behavioral Therapy. Use of CBT-I Coach sleep diaries in Week 0 and Week 6. We measured participant adherence by a count of the number of participants who used the CBT-I Coach at Week 0 (by our definition of use), and the number of participants using the CBT-I Coach at Week 6. Because of the small number of completers and because this is a feasibility study, we provide only descriptive data.
Time Frame: Week 0 (Pre-Intervention) and Week 6 (Post-Intervention)
Population: Those completing enrollment and not withdrawn by study personnel for insomnia were counted at Week 0. The Week 0 outcome measure is the number of participants who used sleep diaries in the CBT-I Coach for 5 or more nights of Week 0. In Week 6 it is the number of participants who used the CBT-I Coach for 5 or more nights during the sixth week.
Measure: Count of Participants; unit: Participants
Arm/Group | WatchPAT and CBT-i Coach App
Number analyzed (Participants) | 11
Participants
  Participants using CBT-I Coach at Baseline | 11
  Participants using CBT-I Coach Week 6 | 9

3. Secondary Outcome: Insomnia Severity Index Score
Description: Validated self-report measure of Insomnia Symptom Severity (ISI). The minimum ISI scale score is 0, the maximum scale score is 28, and higher scores indicate worse insomnia. Because of the small number of completers and because this is a feasibility study, we provide only descriptive data in the form of means (and standard deviation).
Time Frame: Week 0 (Pre-Intervention) and Week 4 (Mid-Intervention) and Week 6 (Post-Intervention)
Population: Those who completed enrollment and were not withdrawn by study personnel for insomnia are considered those who are counted at Week 0.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | WatchPAT and CBT-i Coach App
Number analyzed (Participants) | 11
units on a scale
  Insomnia Severity Score at Baseline | 16.6 (5.6)
  Insomnia Severity Score at Week 4 | 12.4 (4.5)
  Insomnia Severity Score at Week 6 | 12.8 (3.7)

4. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI) Total Score
Description: Validated self-report measure of self-reported sleep quality. The minimum PSQI Total scale score is 0, the maximum scale score is 21 and higher scale scores indicate worse subjective sleep quality. Because of the small number of completers and because this is a feasibility study, we provide only descriptive data in the form of means (and standard deviation).
Time Frame: Week 0 (Pre-Intervention) and Week 4 (Mid-Intervention) and Week 6 (Post-Intervention)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | WatchPAT and CBT-i Coach App
Number analyzed (Participants) | 11
units on a scale
  PSQI Total Score at Baseline | 12.8 (4.6)
  PSQI Total Score at Week 4 | 10.4 (2.7)
  PSQI Total Score at Week 6 | 10.7 (3.3)

5. Secondary Outcome: Functional Outcomes of Sleep Score
Description: Validated self-report short-form (10 item) measure of Functional Outcomes of Sleep-10 (FOSQ-10). The minimum FOSQ score is 5, the maximum score is 20, and higher scores indicate better functioning. Because of the small number of completers and because this is a feasibility study, we provide only descriptive data in the form of means (and standard deviation).
Time Frame: Week 0 (Pre-Intervention) and Week 4 (Mid-Intervention) and Week 6 (Post-Intervention)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | WatchPAT and CBT-i Coach App
Number analyzed (Participants) | 11
units on a scale
  FOSQ Score at Baseline | 13.9 (3.7)
  FOSQ Score at Week 4 | 15.2 (3.8)
  FOSQ Score at Week 6 | 15.4 (2.9)

ADVERSE EVENTS:
Description: We monitored for adverse events only those participants who were eligible and received the intervention.
Arm/Group | WatchPAT and CBT-i Coach App
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes